CLINICAL TRIAL: NCT04381143
Title: ASPIrin in Reducing Events in Dialysis
Brief Title: ASPIrin in Reducing Events in Dialysis ( ASPIRED )
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDPH-CH-2774
Record Dates: First submitted 2020-04-23; First posted 2020-05-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: CKD (Chronic Kidney Disease) Stage 5D
Keywords: Aspirin; Dialysis; End Stage Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Pragmatic designs
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Active Comparator): Aspirin tablet 100mg daily
  Interventions: Drug: Aspirin 100 mg Oral Tablet
- Matching Placebo (Placebo Comparator): Placebo tablet 1 pill daily
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Aspirin 100 mg Oral Tablet — Aspirin 100 mg tablet daily
  Arms: Aspirin
Drug: Matching Placebo — Matching Placebo 1 pill daily
  Arms: Matching Placebo

SUMMARY:
People with kidney failure requiring dialysis have a much higher risk of developing cardiovascular (CV) disease compared with the general population. A cardiac cause accounts for 58% of all deaths in patients with end stage kidney disease (ESKD). At the same time, this population has increased risks of clotting as well as bleeding episodes. While aspirin is known to reduce cardiovascular complications in the general population, evidence to support the use of aspirin in people with ESKD receiving dialysis therapy is currently lacking. The ASPIrin to Reduce Event in Dialysis (ASPIRED) trial will test whether aspirin use in dialysis patients safely improves outcomes compared with no aspirin use.

DETAILED DESCRIPTION:
ASPIRED is an investigator-initiated, multi-center, double-blind, parallel group, event-driven, pragmatic, registry-based randomized controlled trial that will define the value of low dose aspirin (100 mg daily) on cardiovascular events in people with ESKD receiving dialysis.

The study will be conducted using the existing platform of the Chinese peritoneal dialysis (PD) and hemodialysis (HD) Dialysis Registry to screen, recruit and to collect study data as part of patient's routine clinical care during dialysis to improve efficiency and to minimize cost of a clinical trial.

ASPIRED is an event driven trial with an anticipated duration of approximately 5 years.

Randomization will be performed using a web-based system via a pass word protected encrypted website interface.

The study procedure utilizes routine six-monthly clinic visits for study follow-up to increase efficiency and minimize the burden on participants.

The analysis will be based on intention-to-treat principles. An independent Data Safety and Monitoring Board (DSMB) will established to monitor the study for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Incident or prevalent adults (≥18 years old) dialysis patients are included in the Dialysis Registry.
* Commenced on dialysis with the expectation of ongoing maintenance dialysis requirement.
* Willing and able to provide informed consent for this study.

Exclusion Criteria:

* Requirement for any form of antiplatelet agent (aspirin, glycoprotein IIb/IIIa inhibitors etc), or oral anticoagulation (warfarin, NOACs), in the view of the treating physician.
* Contraindication to aspirin, in the view of the treating physician.
* Dialysis requirement due to acute kidney injure with expectation of kidney function recovery.
* History of haemorrhagic stroke or intracranial bleed within 12 months of screening.
* Coagulopathy from any cause.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9000 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with composite of major cardiovascular events (3-point MACE) | From trial initiation to any event first occurrence, up to 5 years.
  A composite of cardiovascular death, myocardial infarction, or ischemic stroke.

SECONDARY OUTCOMES:
Number of Participants with composite of major cardiovascular events plus all-cause death | From trial initiation to any event first occurrence, up to 5 years.
  A composite of cardiovascular death, myocardial infarction, ischemic stroke or all-cause death.
Number of Participants with composite of major cardiovascular events, hospitalised unstable angina (UA) and hospitalised transient ischaemic attack (TIA) | From trial initiation to any event first occurrence, up to 5 years.
  A composite of cardiovascular death, myocardial infarction, ischemic stroke, hospitalised unstable angina (UA) or hospitalised transient ischaemic attack (TIA)
Number of Participants with cardiovascular death | From trial initiation to any event first occurrence, up to 5 years.
  Death due to CV cause.
Number of Participants with Myocardial infarction | From trial initiation to any event first occurrence, up to 5 years.
Number of Participants with ischemic stroke | From trial initiation to any event first occurrence, up to 5 years.
Number of Participants with all-cause death | From trial initiation to any event first occurrence, up to 5 years.
  Death for any reason.
Number of Participants with coronary revascularization | From trial initiation to any event occurrence, up to 5 years.
Number of Participants with fistula or graft thrombosis | From trial initiation to any event occurrence, up to 5 years.
Number of Participants with intracranial haemorrhage | From trial initiation to any event occurrence, up to 5 years.
Number of Participants with peripheral vascular events | From trial initiation to any event occurrence, up to 5 years.
Number of Participants with ischemic events | From trial initiation to any event occurrence, up to 5 years.
  Defined as a composite of myocardial infarction (MI), coronary death, ischemic stroke, or any revascularization procedure (i.e, exclusion of noncoronary cardiac deaths and strokes confirmed to be haemorrhagic).

OTHER OUTCOMES:
Major bleeding | From trial initiation to any event first occurrence, up to 5 years.
  Major bleeding is defined based on modified International Society on Thrombosis and Haemostasis (ISTH) definition, including fatal bleeding, and/or symptomatic bleeding in a critical area or organ, such as intracranial, intra-spinal, intra-ocular, retro-peritoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, or bleeding into a surgical site requiring re-operation, and/or bleeding leading to hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, Study Chair — Guangdong Provincial People's Hospital; Vlado Perkovic, Study Chair — The University of New South Wales Sydney; Muh Geot Wong, Study Director — The George Institute; Wei Chen, Study Director — First Affiliated Hospital, Sun Yat-Sen University; Li Fan, Study Director — Guangdong Provincial People's Hospital; Zhiming Ye, Study Director — Guangdong Provincial People's Hospital
Locations (139):
- China (139):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Shanghang County Hospital, Longyan, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Dongguan Donghua Hospital, Dongguan, Guangdong
  - Dongguan Hospital of Integrative Traditional Chinese and Western Medicine, Dongguan, Guangdong
  - Dongguan Houjie Hospital, Dongguan, Guangdong
  - Dongguan Eighth People's Hospital, Dongguan, Guangdong
  - Dongguan Marina Bay Center Hospital, Dongguan, Guangdong
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Dongguan Songshan Lake Center Hospital, Dongguan, Guangdong
  - Lufeng People's Hospital, Donghai, Guangdong
  - Foshan Gaoming District People's Hospital, Foshan, Guangdong
  - The Second People Hospital of Foshan Nanhai, Foshan, Guangdong
  - Foshan Nanhai District People's Hospital, Foshan, Guangdong
  - Foshan No.1 people's hospital, Foshan, Guangdong
  - Foshan Sanshui People's Hospital, Foshan, Guangdong
  - Foshan Second People's Hospital, Foshan, Guangdong
  - Guangdong Provincial Hospital of Integrative Medicine, Foshan, Guangdong
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Guangzhou Redcross Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine Fangcun Branch (Guangzhou Charity Hospital), Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong Agricultural Reclamation Central Hospital, Guangzhou, Guangdong
  - Guangdong Cliffod Hospital, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Hua Du District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - Panyu District people's hospital of Guangzhou, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guanzhou, Guangdong
  - Heyuan People's Hospital, Heyuan, Guangdong
  - Huizhou First People Hospital, Huizhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - The People's Hospital of Jiangmen, Jiangmen, Guangdong
  - Jiangmen Center hospital, Jiangmen, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Kaiping Center Hospital, Kaiping, Guangdong
  - Lianjiang People's Hospital, Lianjiang, Guangdong
  - Lianping County People's Hospital, Lianping, Guangdong
  - The Fourth Affiliated Hospital of Guangzhou Medical University, Licheng, Guangdong
  - Maoming Hospital of Traditional Chinese Medicine, Maoming, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University Yuedong Hospital, Meizhou, Guangdong
  - Puning People's Hospital, Puning, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Fogang People Hospital, Qingyuan, Guangdong
  - Qingyuan Hospital of Traditional Chinese Medicine, Qingyuan, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - The first Affiliated Hospital of Shantou Medical University, Shantou, Guangdong
  - Shantou Chaonan Minsheng Hospital, Shantou, Guangdong
  - Shanwei People's Hospital, Shanwei, Guangdong
  - Shenshan Medical Center, Memorial Hospital of Sun Yat-sen University, Shanwei, Guangdong
  - Wengyuan People Hospital, Shaoguan, Guangdong
  - Shaoguan First People's Hospital, Shaoguan, Guangdong
  - The First People's Hospital of Shaoguan, Shaoguan, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - The Seventh Affiliated Hospital of Sun Yat-sen, Shenzhen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Baoan People's Hospital, Shenzhen, Guangdong
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - Shenzhen Longhua District People's Hospital, Shenzhen, Guangdong
  - Shenzhen No.2 people's hospital, Shenzhen, Guangdong
  - The Eighth Affiliated Hospital of Sun Yat-sen University (Futian, Shenzhen), Shenzhen, Guangdong
  - ShunDe Hospital Guangzhou University of Chinese Medicine, Shunde, Guangdong
  - The Eighth Affiliated Hospital of Southern Medical University, The First People's Hospital of Shunde, Shunde, Guangdong
  - Nanxiong People Hospital, Xiongzhou, Guangdong
  - People's Hospital of Yangdong District Yangjiang City, Yangjiang, Guangdong
  - Yangjiang Hospital of Traditional Chinese Medicine, Yangjiang, Guangdong
  - Yangjiang People's Hospital, Yangjiang, Guangdong
  - People Hospital of Yingde City Guangdong Province, Yingcheng, Guangdong
  - Yunfu People's Hospital, Yunfu, Guangdong
  - The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Central People's Hospital of Zhanjiang, Zhanjiang, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University Zhaoqing Hospital, Zhaoqing, Guangdong
  - Zhaoqing first people's hospital, Zhaoqing, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - Zhongshan Traditional Chinese Hospital, Zhongshan, Guangdong
  - Zhongshan Xiaolan People's Hospital, Zhongshan, Guangdong
  - Jinwan Center Hospital of Zhuhai, Zhuhai, Guangdong
  - The fifth affiliated hospital of sun yat-sen university, Zhuhai, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - Shantou Central Hospital, Shantou, Guanggong
  - The Affiliated Hospital of Youjiang Ethnic Medicine College, Baise City, Guangxi
  - The first affiliated hospital of Guangxi Medical University, Nanning, Guangxi
  - Anshun Xixiu District People's Hispital, Anshun, Guizhou
  - China Guihang 302 Hospital, Anshun, Guizhou
  - Anshun People Hospital, Anshun, Guizhou
  - Guizhou Province Peple's Hospital, Guiyang, Guizhou
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - Xinyang Central Hospital, Xinyang, Henan
  - Huangshi Central Hospital, Huangshi, Hubei
  - Jingmen Central Hospital, Jingmen, Hubei
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Wuhan Puren Hospital, Wuhan, Hubei
  - The First People's Hospital of Jiangxia District, Wuhan City, Wuhan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - The Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of Huazhong Science and Technology University, Wuhan, Hubei
  - Wuhan No.1 People's Hospital, Wuhan, Hubei
  - Yichang central people's hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Nantong Haimen People's Hospital, Nantong, Jiangsu
  - Xuzhou Mining Group General Hospital, Xuzhou, Jiangsu
  - Subei People's Hospital, Yangzhou, Jiangsu
  - Ganzhou Municiple Hospital, Ganzhou, Jiangxi
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - Jiujiang No.1people's Hospital, Jiujiang, Jiangxi
  - Jiangxi Province Peple's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The Second Affiliated Hospital of Xi'an Jiaotong University (Xibei Hospital), Xi’an, Shanxi
  - The First Affiliated Hospital of Air Force Military Medical University, Xi’an, Shanxi
  - Sichuan Province People's Hospital, Chengdu, Sichuan
  - Jiashi County People's Hospital, Kashgar, Xinjiang
  - Shache County People's Hospital, Kashgar, Xinjiang
  - The First People's Hospital of Kashi Prefecture, Kashgar, Xinjiang
  - The Second People's Hospital of Kashi Prefecture, Kashgar, Xinjiang
  - The First Affiliated Hospital of Shihezi University Medical College, Shihezi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The People's hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Fengqing People's Hospital of Yunnan Province, Lincang, Yunnan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Lishui City Center Hospital, Lishui, Zhejiang
  - Zhoushan Hospital, Zhoushan, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data that supports the results will be shared following publication. Any sub-study analysis and publication will have to be reviewed and approved by the Trial Steering Committee, local Ethics and Regulatory requirements.